CLINICAL TRIAL: NCT05642234
Title: Comparison of Skin - Epidural and Intervertebral Distances Measured by Ultrasonography in Sitting and Rider Position
Brief Title: Comparison of Skin - Epidural and Intervertebral Distances in Sitting and Rider Position
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nazim Ufuk Turhaner, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 367794
Record Dates: First submitted 2022-11-28; First posted 2022-12-08 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Anesthesia, Epidural; Analgesia, Epidural; Ultrasound Imaging
Keywords: Epidural anesthesia; Rider position; İntervertebral distance; Skin-epidural distance
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Epidural Ultrasonography — In this study, we measured the intervertebral distance and skin-epidural distance with the help of ultrasonography in the thoracic and lumbar regions in sitting and rider positions.

SUMMARY:
Epidural anesthesia/analgesia can be performed under various positions. In this study, the investigators aimed to compare the intervertebral and skin-epidural distances in "the sitting" and "rider" positions with the help of ultrasonography

DETAILED DESCRIPTION:
Complication rates in epidural intervention, which can be used for both intraoperative and postoperative analgesia are higher than peripheral blocks, especially in open abdominal surgeries. In epidural intervention, correct determination of patient position, puncture site and the distance from the skin to the epidural area (skin - epidural distance) is very important in terms of preventing complications. The location of the point where the epidural intervention will be made is aimed to be determined using the anatomical surface markings in the blind technique. However, anatomical surface markings are unreliable in pregnant or obese patients and patients with anatomical variants. The use of pre-procedure ultrasonography allows obtaining information such as midline and baseline determination, skin-epidural distance measurement, increasing the success of the intervention.

The most preferred positions for epidural interventions are sitting and lateral decubitus positions. Many modifications of these positions also exist. The rider position is used in a few centers in and out of Turkey, but there is only one clinical study related to the position.

ELIGIBILITY:
Inclusion Criteria:

• ASA (American Society of Anesthesiologists) classification I-III

Exclusion Criteria:

* Prior spinal surgery
* Spinal deformity
* Recent spinal and head trauma
* Infection in the area to be measured
* Severe hypovolemia
* Severe edema
* severe abdominal distention
* Severe pain
* Difficulty in cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is carried out in patients over 18 years of age who will undergo abdominal surgery, with ASA (American Society of Anesthesiologists) classification I-III.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Intervertebral distance | 5 minutes
  Comparison of intervertebral distance measurements with the help of ultrasonography in the thoracic and lumbar regions in sitting and rider positions.
Skin - epidural distance | 5 minutes
  Comparison of skin - epidural distance measurements with the help of ultrasonography in the thoracic and lumbar regions in sitting and rider positions.

CONTACTS AND LOCATIONS:
Overall Officials: Safak Emre Erbabacan, MD, Study Chair — Istanbul University - Cerrahpasa; Fatis Altındas, Prof., Study Director — Istanbul University - Cerrahpasa; Cigdem Akyol Beyoglu, Assoc. Prof., Study Director — Istanbul University - Cerrahpasa; Aylin Nizamoglu, Assoc. Prof., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We will share information about gender, age, height, body weight, ASA class, diagnosis, surgery, thoracic and lumbar intervertebral and skin-epidural distances measured in the rider and sitting positions

REFERENCES:
- [Background] Korkmaz Toker M, Altiparmak B, Uysal AI, Turan M, Gumus Demirbilek S. Rider sitting position widens lumbar intervertebral distance: a prospective observational study. Braz J Anesthesiol. 2023 Nov-Dec;73(6):758-763. doi: 10.1016/j.bjane.2021.03.010. Epub 2021 Apr 19. PMID 33887338
- [Background] Sahin T, Balaban O, Sahin L, Solak M, Toker K. A randomized controlled trial of preinsertion ultrasound guidance for spinal anaesthesia in pregnancy: outcomes among obese and lean parturients: ultrasound for spinal anesthesia in pregnancy. J Anesth. 2014 Jun;28(3):413-9. doi: 10.1007/s00540-013-1726-1. Epub 2013 Oct 20. PMID 24141882
- [Background] Sahin T, Balaban O. Lumbar Ultrasonography for Obstetric Neuraxial Blocks: Sonoanatomy and Literature Review. Turk J Anaesthesiol Reanim. 2018 Aug;46(4):257-267. doi: 10.5152/TJAR.2018.90277. Epub 2018 Aug 1. PMID 30140531
- [Background] Khemka R, Rastogi S, Desai N, Chakraborty A, Sinha S. Comparison of ultrasound imaging in transverse median and parasagittal oblique planes for thoracic epidurals: A pilot study. Indian J Anaesth. 2016 Jun;60(6):377-81. doi: 10.4103/0019-5049.183398. PMID 27330197
- [Background] Soltani Mohammadi S, Piri M, Khajehnasiri A. Comparing Three Different Modified Sitting Positions for Ease of Spinal Needle Insertion in Patients Undergoing Spinal Anesthesia. Anesth Pain Med. 2017 Oct 23;7(5):e55932. doi: 10.5812/aapm.55932. eCollection 2017 Oct. PMID 29696117
- [Background] Soltani Mohammadi S, Hassani M, Marashi SM. Comparing the squatting position and traditional sitting position for ease of spinal needle placement: a randomized clinical trial. Anesth Pain Med. 2014 Apr 5;4(2):e13969. doi: 10.5812/aapm.13969. eCollection 2014 May. PMID 24790901